CLINICAL TRIAL: NCT01633970
Title: A Phase Ib Study of the Safety and Pharmacology of Atezolizumab (Anti-PD-L1 Antibody) Administered With Bevacizumab and/or Chemotherapy in Patients With Advanced Solid Tumors
Brief Title: A Study of Atezolizumab Administered in Combination With Bevacizumab and/or With Chemotherapy in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP28328; 2012-001422-10 (EudraCT Number)
Record Dates: First submitted 2012-06-22; First posted 2012-07-06 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Fluorouracil; atezolizumab; Bevacizumab; Carboplatin; Leucovorin; 130-nm albumin-bound paclitaxel; Oxaliplatin; Paclitaxel; Pemetrexed

ARMS (6):
- A: Atezolizumab + Bevacizumab (Experimental): Participants will receive atezolizumab 10 milligrams per kilogram (mg/kg) intravenous (IV) infusion (or a selected dose level not to exceed the single agent MTD or MAD determined in Study PCD4989g) with bevacizumab 15 mg/kg every 3 weeks (q3w). After establishment of MTD or MAD, participants will receive bevacizumab 15 mg/kg IV infusion on Day 1 of Cycle 1 followed by atezolizumab 1200 mg IV infusion q3w after Days 5-7 and then atezolizumab 1200 mg q3w and bevacizumab 15 mg/kg q3w on Day 1 of all subsequent cycles until disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- B: Atezolizumab + Bevacizumab + FOLFOX (Experimental): Participants will receive FOLFOX IV infusion (oxaliplatin [85 milligrams per square meter {mg/m^2}], leucovorin [400 mg/m^2], 5-FU [400 mg/m^2]) on Day 1 of Cycle 1 and then atezolizumab 800 mg IV infusion every 2 weeks (q2w), bevacizumab 10 mg/kg IV infusion q3w and FOLFOX q2w on Day 1 of all subsequent cycles as per institutional guidelines until disease progression or unacceptable toxicity.
  Interventions: Drug: 5-FU; Drug: Atezolizumab; Drug: Bevacizumab; Drug: Leucovorin; Drug: Oxaliplatin
- C: Atezolizumab + Carboplatin + Paclitaxel (Experimental): Participants will receive atezolizumab 1200 mg IV infusion q3w in combination with paclitaxel 200 mg/m^2 IV infusion q3w and then carboplatin IV q3w (on Day 1 of every 3-week cycle) to achieve an initial target area under the curve (AUC) of 6 milligrams per milliliter*minute (mg/mL*min) until disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Paclitaxel
- D: Atezolizumab + Carboplatin + Pemetrexed (Experimental): Participants will receive atezolizumab 1200 mg IV infusion q3w in combination with premetrexed 500 mg/m^2 IV infusion q3w and then carboplatin IV q3w (on Day 1 of every 3-week cycle) to achieve an initial target AUC of 6 mg/mL*min until disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Pemetrexed
- E: Atezolizumab + Carboplatin + Nab-paclitaxel (Experimental): Participants will receive atezolizumab 1200 mg IV infusion q3w (on Day 1 of every 3-week cycle) in combination with nab-paclitaxel 100 mg/m^2 IV infusion once weekly (qw) (on Days 1, 8 and 15 of every 3-week cycle) and then carboplatin IV infusion q3w (on Day 1 of every 3-week cycle) to achieve an initial target AUC of 6 mg/mL*min until disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Nab-paclitaxel
- F: Atezolizumab + Nab-paclitaxel (Experimental): Participants will receive atezolizumab 800 mg IV infusion q2w (Days 1 and 15) in combination with nab-paclitaxel 125 mg/m^2 IV infusion qw (on Days 1, 8 and 15 of every 3-week cycle) until disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: 5-FU — Participants will receive 5-FU 400 mg/m^2 IV q2w.
  Arms: B: Atezolizumab + Bevacizumab + FOLFOX
Drug: Atezolizumab — Participants will receive IV atezolizumab (800 mg q2w or 1200 mg q3w) q3w.
  Other Names: MPDL3280A
Drug: Bevacizumab — Participants will receive bevacizumab 10 mg/kg or 15 mg/kg IV q3w.
  Other Names: Avastin
  Arms: A: Atezolizumab + Bevacizumab; B: Atezolizumab + Bevacizumab + FOLFOX
Drug: Carboplatin — Participants will receive carboplatin IV q3w with target AUC of 6 mg/mL.
  Arms: C: Atezolizumab + Carboplatin + Paclitaxel; D: Atezolizumab + Carboplatin + Pemetrexed; E: Atezolizumab + Carboplatin + Nab-paclitaxel
Drug: Leucovorin — Participants will receive leucovorin 400 mg/m^2 IV q2w.
  Arms: B: Atezolizumab + Bevacizumab + FOLFOX
Drug: Nab-paclitaxel — Participants will receive nab-paclitaxel 100 mg/m^2 IV qw.
  Arms: E: Atezolizumab + Carboplatin + Nab-paclitaxel; F: Atezolizumab + Nab-paclitaxel
Drug: Oxaliplatin — Participants will receive oxaliplatin 85 mg/m^2 IV q2w.
  Arms: B: Atezolizumab + Bevacizumab + FOLFOX
Drug: Paclitaxel — Participants will receive paclitaxel 200 mg/m^2 IV q3w.
  Arms: C: Atezolizumab + Carboplatin + Paclitaxel
Drug: Pemetrexed — Participants will receive pemetrexed 500 mg/m^2 IV q3w.
  Arms: D: Atezolizumab + Carboplatin + Pemetrexed

SUMMARY:
This open-label, Phase Ib study that has six treatment arms is designed to assess the safety, pharmacology and preliminary efficacy of atezolizumab (MPDL3280A; an engineered anti-programmed death-ligand 1 [PDL1] antibody) administered with bevacizumab (Arm A) and with bevacizumab plus oxaliplatin, leucovorin, and 5-fluorouracil (5-FU) (FOLFOX) (Arm B), with carboplatin and paclitaxel (Arm C), with carboplatin and pemetrexed (Arm D), with carboplatin and nab-paclitaxel (Arm E), and with nab-paclitaxel (Arm F) in participants with locally advanced or metastatic solid tumors. The study includes dose escalation cohort for establishing the maximum tolerated dose (MTD) or maximum administered dose (MAD) and then expansion cohort will be initiated based on a selected dose level at or below the MTD or MAD.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Histologically or cytologically documented advanced solid tumors
* Adequate hematologic and end organ function
* Measurable disease by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Resolution of any acute, clinically significant treatment-related toxicity from prior therapy to Grade less than or equal to (</=) 1 prior to study entry, with the exception of alopecia

Eligible Tumor Types:

Arm A Escalation Cohorts and Arms A and B Biopsy Cohort (Cutaneous/Subcutaneous Lesions)

* Histologically or cytologically documented, incurable or metastatic solid malignancy that has failed all available or acceptable standard therapy for which the participant is eligible Arm A and B Safety Expansion Cohorts, Arm B Escalation Cohorts, and Arm B Biopsy Cohort (Liver Lesions)
* Histologically or cytologically confirmed metastatic colorectal cancer (mCRC). Participants in the Arm A Safety Expansion Cohort must have mCRC for which established therapies have proved ineffective or intolerable. Participants with malignancies other than mCRC within 5 years prior to Day 1 (except for those with a negligible risk of metastasis or death, such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) are not eligible.

Arm A renal cell carcinoma (RCC) Cohort:

- Histologically or cytologically confirmed advanced or metastatic RCC with a clear cell component.

Arm A Tumor Type-Specific Cohort:

Gastric Cancer:

- Histologically or cytologically confirmed locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction for which established therapies have proved ineffective or intolerable. The decision may be made to restrict enrollment to participants with a specified tumor PD-L1 status (e.g., immunohistochemistry [IHC] status 0/1 or 2/3)

Ovarian Cancer:

- Measurable/assessable ovarian cancer (defined as epithelial ovarian, fallopian tube, or primary peritoneal cancer) that has progressed less than (<) 6 months after completing platinum-based therapy. The following histological types are eligible: Adenocarcinoma NOS, clear cell adenocarcinoma, endometriod adenocarcinoma, malignant Brenner's tumour, mixed epithelial carcinoma, mucinous adenocarcinoma, serous adenocarcinoma, transitional cell carcinoma, undifferentiated carcinoma

Bladder Cancer:

* Histologically or cytologically documented locally advanced (T4b, any N; or any T, N 2-3) or metastatic (M1, Stage IV) transitional cell carcinoma of the urothelium (including renal pelvis, ureters, urinary bladder, urethra)
* Participants with mixed histologies are required to have a dominant transitional cell pattern
* Locally advanced bladder cancer must be inoperable based on involvement of pelvic sidewall or adjacent viscera (clinical stage T4b) or bulky nodal metastasis (N2-N3)
* Disease progression during or following treatment with at least one platinum-containing regimen (e.g., GC, MVAC, CarboGem, etc.) for inoperable locally advanced or metastatic urothelial carcinoma or disease recurrence

Cervical Cancer:

* Persistent or recurrent squamous cell carcinoma of the cervix (including adenosquamous tumors)

Arms C, D, and E Cohorts:

- Histologically or cytologically documented Stage IIIB (not eligible for definitive chemoradiotherapy), Stage IV, or recurrent non-small cell lung cancer (NSCLC)

Arm F Cohort:

* Histologically confirmed estrogen receptor (ER)-, progesterone receptor (PR)-, and human epidermal growth factor receptor (HER)-negative (triple-negative) adenocarcinoma of the breast that has been treated with systemic cytotoxic therapy. Locally recurrent disease must not be amenable to resection with curative intent
* Participants with tumors amenable to excisional, punch, or core needle biopsy are eligible for a separate biopsy expansion cohort

Tumor molecular status:

Arm A safety expansion cohort

- Up to 10 participants with CRC and high microsatellite instability (MSI-H) may be enrolled

Exclusion Criteria:

General Exclusions

* Any approved anti-cancer therapy, including chemotherapy, hormonal therapy, radiotherapy, or herbal therapy intended as anti-cancer therapy, within 3 weeks prior to initiation of study treatment; the following are allowed: hormonal therapy with gonadotropin-releasing hormone agonists or antagonists for prostate cancer, hormone-replacement therapy, and palliative radiotherapy for bone metastases greater than (>) 2 weeks prior to Day 1
* Bisphosphonate therapy for symptomatic hypercalcemia
* Known clinically significant liver disease
* Known primary central nervous (CNS) malignancy or active CNS metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control)
* Pregnant or lactating women
* Known hypersensitivity to Chinese hamster ovary cell products or any component of the atezolizumab formulation
* History of autoimmune disease, idiopathic pulmonary fibrosis, human immunodeficiency virus (HIV), hepatitis B or C infection; history of hepatitis B is allowed if infection has resolved (absence of hepatitis B surface antigen [HBsAg])
* Severe infections within 4 weeks prior to Day 1, or signs or symptoms of significant infection within 2 weeks prior to Day 1
* Received oral or IV antibiotics within 2 weeks prior to Cycle 1 Day 1
* History of myocardial infarction, unstable angina stroke or transient ischemic attack within 6 months prior to Day 1
* Administration of a live, attenuated vaccine within 4 weeks before Day 1 or anticipation that such a live attenuated vaccine will be required during the study Bevacizumab-Specific Exclusions (Arms A and B) Exclusion Criteria Unique to Arm A RCC Cohort
* Any prior systemic treatment (including tyrosine kinase inhibitors, antibody therapy, immunotherapy, chemotherapy, hormonal therapy, or investigational therapy) for RCC. All treatments, neo-adjuvant, adjuvant, or for locally advanced or metastatic RCC are not permitted

Arm A Tumor Type-Specific Cohort:

Gastric Cancer:

- Prior approved or experimental anti-vascular endothelial growth factor or its receptor (VEGF/VEGFR) therapy (including, for example, bevacizumab or nintedanib). The decision may be made to allocate a specified number of slots to participants who have received prior anti-VEGF/VEGFR therapy

Ovarian Cancer:

* Refractory disease
* History of bowel obstruction
* >2 prior anticancer regimens
* Prior approved or experimental anti-VEGF/VEGFR therapy (including, for example, bevacizumab or nintedanib)

Cervical Cancer:

- > 2 prior cytotoxic regimens, not including prior cisplatin-based chemotherapy concomitantly administered with primary pelvic radiation

Exclusion Criteria Unique to Arm B:

* Prior treatment with an oxaliplatin-containing regimen. Oxaliplatin >12 months prior to the diagnosis of metastatic disease is permitted.
* Known dihydropyrimidine dehydrogenase deficiency or thymidylate synthase gene polymorphism predisposing the participant for 5-FU toxicity

Exclusion Criteria Unique to Arms C, D, and E:

* Prior chemotherapy for locally advanced or metastatic NSCLC
* For participants who received prior adjuvant/neo-adjuvant chemotherapy or chemoradiation for NSCLC, a treatment-free interval >6 months between the last treatment administration and the date of recurrence in required
* Participants with a known epidermal growth factor receptor (EGFR) sensitizing mutation must have experienced disease progression during or after treatment with an approved EGFR tyrosine kinase inhibitor
* Participants with a known anaplastic lymphoma kinase (ALK) fusion oncogene must have experienced disease progression during or after treatment with crizotinib
* For Arm D (carboplatin + pemetrexed), squamous cell histology or evidence of mixed NSCLC histology with a predominance of the squamous cell type
* For Arm D (carboplatin + pemetrexed), inability to discontinue treatment with non-steroidal anti-inflammatory drugs (NSAIDs) for 5 days

Exclusion Criteria Unique to Arm F:

* Prior therapy with more than two cytotoxic regimens for metastatic or locally advanced triple-negative breast cancer (TNBC)
* Treatment with a taxane-containing regimen within 6 months before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-07-11 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Atezolizumab Dose | Days 1-21 of Cycle 1 (Cycle length = 21 days) for Arms A, C, D and E and the 28 days following the first administration of atezolizumab in Arm B
Percentage of Participants With Adverse Events | From Baseline up to 90 days after last dose of study drug or until initiation of another anti-cancer therapy (up to approximately 5 years)
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | Days 1-21 of Cycle 1 (Cycle length = 21 days) for Arms A, C, D and E and the 28 days following the first administration of atezolizumab in Arm B

SECONDARY OUTCOMES:
Duration of Objective Response According to RECIST v1.1 | From Baseline until death or disease progression, whichever occurs first (up to approximately 5 years)
Duration of Objective Response According to irRC | From Baseline until death or disease progression, whichever occurs first (up to approximately 5 years)
Progression-Free Survival According to RECIST v1.1 | From treatment initiation until documented disease progression or death from any cause, whichever occurs first (up to approximately 5 years)
Progression-Free Survival According to irRC | From treatment initiation until documented disease progression or death from any cause, whichever occurs first (up to approximately 5 years)
Pharmacokinetics: Area Under the Serum Concentration-Time Curve (AUC) of Atezolizumab | Pre-infusion (0 hour [hr]) on Cycle 1 Day 1 (cycle length = 21 or 14 days) up to approximately 5 years (detailed timeframe is provided in outcome measure description)
Pharmacokinetics: Maximum Serum Concentration (Cmax) of Atezolizumab | Pre-infusion (0 hr) on Cycle 1 Day 1 (cycle length = 21 or 14 days) up to approximately 5 years (detailed timeframe is provided in outcome measure description)
Minimum Serum Concentration (Cmin) of Atezolizumab | Pre-infusion (0 hr) on Cycle 1 Day 1 (cycle length = 21 or 14 days) up to approximately 5 years (detailed timeframe is provided in outcome measure description)
Percentage of Participants With Best Overall Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | From Baseline until death or disease progression, whichever occurs first (up to approximately 5 years)
Percentage of Participants With Best Overall Response According to Immune-Related Response Criteria (irRC) | From Baseline until death or disease progression, whichever occurs first (up to approximately 5 years)
Percentage of Participants With Objective Response (Complete Response + Partial Response) According to RECIST v1.1 | From Baseline until death or disease progression, whichever occurs first (up to approximately 5 years)
Percentage of Participants With Objective Response (Complete Response + Partial Response) According to irRC | From Baseline until death or disease progression, whichever occurs first (up to approximately 5 years)
Pharmacokinetics: Clearance of Atezolizumab | Pre-infusion (0 hr) on Cycle 1 Day 1 (cycle length = 21 or 14 days) up to approximately 5 years (detailed timeframe is provided in outcome measure description)
Pharmacokinetics: Volume of Distribution of Atezolizumab | Pre-infusion (0 hr) on Cycle 1 Day 1 (cycle length = 21 or 14 days) up to approximately 5 years (detailed timeframe is provided in outcome measure description)
Pharmacokinetics: Accumulation Ratio of Atezolizumab | Pre-infusion (0 hr) on Cycle 1 Day 1 (cycle length = 21 or 14 days) up to approximately 5 years (detailed timeframe is provided in outcome measure description)
Pharmacokinetics: Half-Life of Atezolizumab | Pre-infusion (0 hr) on Cycle 1 Day 1 (cycle length = 21 or 14 days) up to approximately 5 years (detailed timeframe is provided in outcome measure description)
Pharmacokinetics: Cmax of Bevacizumab | Pre-infusion (0 hr), 0.5 hrs after EOI (infusion duration=90 min) on Day 1 Cycles 1 & 3 (each cycle = 21 days); EOT; every 30 days (for up to 120 days) after EOT until death or withdrawal or study closure (up to approximately 5 years)
Pharmacokinetics: Cmin of Bevacizumab | Pre-infusion (0 hr), 0.5 hrs after EOI (infusion duration=90 min) on Day 1 Cycles 1 & 3 (each cycle = 21 days); EOT; every 30 days (for up to 120 days) after EOT until death or withdrawal or study closure (up to approximately 5 years)
Maximum Plasma Concentration of 5-FU | Pre- infusion (0 hr) on Day 1 Cycle 1; end of 5-FU bolus and 2 and 12-24 hrs after end of 5-FU bolus (infusion duration = 46 hrs) on Day 1 of Cycles 1 and 3 (each cycle=14 days)
Pharmacokinetics: Maximum Plasma Concentration of Oxaliplatin | Pre-infusion (0 hr) on Day 1 Cycle 1; 5-10 min before end of oxaliplatin infusion (infusion duration = 120 min) and 2 and 12-24 hrs after end of 5-FU bolus (infusion duration = 46 hrs) on Day 1 of Cycles 1 and 3 (each cycle=14 days)
Pharmacokinetics: Maximum Plasma Concentration of Carboplatin | Pre-infusion (0 hr), 5-10 min before and 1 hr after carboplatin EOI (infusion duration=15-30 min),24 hr after atezolizumab EOI (infusion duration=90 min)on Day 1 Cycle 1; 5-10 min before and 1 hr after carboplatin EOI Day 1 Cycle 3 (each cycle=21 days)
Maximum Plasma Concentration of Paclitaxel | Pre-infusion (0 hr), 5-10 min before and 1 hr after paclitaxel EOI (infusion duration=180 min), 24 hr after atezolizumab EOI (infusion duration=90 min) on Day 1 Cycle 1; 5-10 min before and 1 hr after paclitaxel EOI on Day 1 Cycle 3 (each cycle=21 days)
Pharmacokinetics: Maximum Plasma Concentration of Pemetrexed | Pre-infusion (0 hr), 5-10 min before and 1 hr after pemetrexed EOI (infusion duration=10 min), 24 hr after atezolizumab EOI (infusion duration=90 min) on Day 1 Cycle 1; 5-10 min before and 1 hr after pemetrexed EOI on Day 1 Cycle 3 (each cycle = 21 days)
Maximum Plasma Concentration of Nab-Paclitaxel (Total Paclitaxel) | Pre-infusion (0 hr), 5-10 min before and 1 hr after nab-paclitaxel EOI (infusion duration=30 min) on Day 1 of Cycles 1 and 3; 24 hr after atezolizumab EOI (infusion duration=90 min) on Day 1 Cycle 1 (each cycle=7 days)
Number of Cycles of Each Component of Treatment Administer | From Baseline up to approximately 5 years
Dose Intensity of Each Component of Treatment Administer | From Baseline up to approximately 5 years
Overall Survival (OS) | From first dose of study treatment until death from any cause (up to approximately 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (11):
- United States (11):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Uni of Chicago, Chicago, Illinois
  - Massachusetts General Hospital., Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Dana Farber Can Ins, Boston, Massachusetts
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Carolina BioOncology Institute; Can Therapy & Res Ctr, Huntersville, North Carolina
  - Sarah Cannon Research Inst., Nashville, Tennessee

REFERENCES:
- [Derived] Adams S, Diamond JR, Hamilton E, Pohlmann PR, Tolaney SM, Chang CW, Zhang W, Iizuka K, Foster PG, Molinero L, Funke R, Powderly J. Atezolizumab Plus nab-Paclitaxel in the Treatment of Metastatic Triple-Negative Breast Cancer With 2-Year Survival Follow-up: A Phase 1b Clinical Trial. JAMA Oncol. 2019 Mar 1;5(3):334-342. doi: 10.1001/jamaoncol.2018.5152. PMID 30347025
- [Derived] Liu SV, Camidge DR, Gettinger SN, Giaccone G, Heist RS, Hodi FS, Ready NE, Zhang W, Wallin J, Funke R, Waterkamp D, Foster P, Iizuka K, Powderly J. Long-term survival follow-up of atezolizumab in combination with platinum-based doublet chemotherapy in patients with advanced non-small-cell lung cancer. Eur J Cancer. 2018 Sep;101:114-122. doi: 10.1016/j.ejca.2018.06.033. Epub 2018 Jul 24. PMID 30053670